CLINICAL TRIAL: NCT05870319
Title: A Randomized, Open-Label, Multicenter Phase 3 Study to Evaluate SKB264 Monotherapy Versus Pemetrexed in Combination With Platinum in Patients With Locally Advanced or Metastatic Non-squamous Non-small Cell Lung Cancer With EGFR Mutation Who Have Failed to Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor (EGFR-TKI) Therapy
Brief Title: A Phase III Study of SKB264 for EGFR Mutant NSCLC Patients
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sichuan Kelun-Biotech Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sichuan Kelun Pharmaceutical Research Institute Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SKB264-Ⅲ-09
Record Dates: First submitted 2023-04-18; First posted 2023-05-23 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Carboplatin; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SKB264 by IV infusion on Days 1 and 15 of each 4-week cycle; (Experimental)
  Interventions: Drug: SKB264
- pemetrexed+ carboplatin or on Day 1 of each 3-week cycle, with 4 cycles chemo (Active Comparator)
  Interventions: Drug: Pemetrexed; Drug: Carboplatin; Drug: Cisplatin

INTERVENTIONS:
Drug: SKB264 — intravenous (IV) infusion (Q2W)
  Arms: SKB264 by IV infusion on Days 1 and 15 of each 4-week cycle;
Drug: Pemetrexed — 500 mg/m2 intravenous (IV) infusion (Q3W)
  Arms: pemetrexed+ carboplatin or on Day 1 of each 3-week cycle, with 4 cycles chemo
Drug: Carboplatin — AUC 5 intravenous (IV) infusion (Q3W) 4cycles
  Arms: pemetrexed+ carboplatin or on Day 1 of each 3-week cycle, with 4 cycles chemo
Drug: Cisplatin — 75 mg/m2 intravenous (IV) infusion (Q3W) 4cycles
  Arms: pemetrexed+ carboplatin or on Day 1 of each 3-week cycle, with 4 cycles chemo

SUMMARY:
This is a randomized, open-label, multicenter Phase 3 clinical study to evaluate SKB264 monotherapy versus pemetrexed in combination with platinum in subjects with locally advanced or metastatic non-squamous NSCLC with EGFR mutation who have failed to EGFR-TKI therapy.

DETAILED DESCRIPTION:
This is a randomized, open-label, multicenter Phase 3 clinical study to evaluate SKB264 monotherapy versus pemetrexed in combination with platinum in subjects with locally advanced or metastatic non-squamous NSCLC with EGFR mutation who have failed to EGFR-TKI therapy. The primary objective is to compare the efficacy and safety of SKB264 monotherapy versus pemetrexed in combination with platinum in patients with locally advanced or metastatic non-squamous NSCLC with EGFR mutation who have failed to EGFR-TKI therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged ≥18 to ≤75 years at the time of signing the ICF;
2. Histologically or cytologically confirmed non-squamous NSCLC and locally advanced (stage IIIB/IIIC) or metastatic (Stage IV) non-squamous NSCLC not amenable to radical surgery and/or radical concurrent/sequential chemoradiotherapy;
3. EGFR-sensitive mutations;
4. Failure of prior EGFR-TKI therapy;
5. At least one measurable target lesion per RECIST 1.1 as assessed by the investigator;
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
7. Expected survival ≥12 weeks;
8. Adequate organ and bone marrow function;
9. Female subjects of childbearing potential and male subjects with partners of childbearing potential who use effective medical contraception from the time of signing the informed consent form until 6 months after the last dose;
10. Subjects voluntarily participate in the study, sign the ICF, and will be able to comply with the protocol-specified visits and relevant procedures

Exclusion Criteria:

1. Histologically or cytologically confirmed presence of small cell lung cancer, neuroendocrine carcinoma, and carcinosarcoma components or squamous cell carcinoma components of more than 10%;
2. Other malignancies within 3 years prior to the first dose;
3. History of (noninfectious) interstitial lung disease (ILD)/noninfectious pneumonitis requiring steroid therapy and current ILD/noninfectious pneumonitis;
4. Subjects with active chronic inflammatory bowel disease, GI tract obstruction, severe ulcers, perforation gastrointestinal, abdominal abscess, or acute GI tract bleed;
5. Toxicities from prior anti-tumor therapy not recovering to ≤ Grade 1 (per NCI CTCAE 5.0) or to the level specified in the eligibility criteria;
6. Subjects with human immunodeficiency virus (HIV) test positive or history of acquired immunodeficiency syndrome (AIDS); known active syphilis infection;
7. Prior TROP2-targeted therapy;
8. Prior treatment with any drug therapy targeting topoisomerase I inhibitor, including antibody-drug conjugates (ADCs);
9. Major surgery within 4 weeks prior to the first dose or expected to require major surgery during the study;
10. Subjects who have received live vaccines within 30 days prior to the first dose, or are scheduled to receive live vaccines during the study;
11. Pregnant or lactating women;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2023-06-26 (Actual); Primary Completion 2024-07-11 (Actual); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From baseline until disease progression, death, or other protocol defined reason,up to approximately 36 months
  PFS assessed by BIRC per RECIST 1.1

SECONDARY OUTCOMES:
Overall survival (OS) | From the date of randomization to the date of death due to any cause. Up to 2 years.
  Overall survival (OS)
Progression-free survival (PFS) | From baseline until disease progression, death, or other protocol defined reason,up to approximately 36 months
  PFS assessed by the investigator per RECIST 1.1
Objective response rate(ORR) | Up to 2 years
  ORR assessed by the investigator and BIRC per RECIST 1.1
Disease control rate(DCR) | Up to 2 years
  DCR assessed by the investigator and BIRC per RECIST 1.1
Duration of response(DOR) | From baseline until disease progression, death, or other protocol defined reason, up to approximately 36 months
  DOR assessed by the investigator and BIRC per RECIST 1.1
Time to response(TTR) | Up to 2 years
  TTR assessed by the investigator and BIRC per RECIST 1.1
AEs and SAEs | AEs should be observed and recorded from signing the ICF until 30 days after the last dose. AEs occurring 30 days after the last dose are not required to be actively collected by the investigator.
  Incidence and severity of AEs and SAEs (per CTCAE 5.0), and clinically significant abnormal laboratory findings
Mean change from baseline in the European Organisation for Research and Treatment of Cancer (EORTC) 30-item core quality-of-life questionnaire (QLQ-C30） | Up to 2 years
  To assess the impact of SKB264 on disease related symptoms and health related quality of life (HRQoL) in this patient population.
Mean change from baseline in the European Organisation for Research and Treatment of Cancer (EORTC) complementary 13-item quality-of-life questionnaire - lung cancer symptoms questionnaire (QLQ-LC13) | Up to 2 years
  To assess the impact of SKB264 on disease related symptoms and health related quality of life (HRQoL) in this patient population

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Fang W, Wu L, Meng X, Yao Y, Zuo W, Yao W, Xie Y, Zhang Y, Cui J, Zhang Y, Li X, Zhuang W, Fang J, Wang Q, Jiang W, Li K, Bai Y, Luo Y, Ma F, Yu Y, Zheng W, Liu Z, Yang B, Ma R, Fang Y, Yang R, Jiang L, Hu J, Yang J, Diao Y, Jin X, Ge J, Yang Y, Zhang L. Sacituzumab Tirumotecan in EGFR-TKI-Resistant, EGFR-Mutated Advanced NSCLC. N Engl J Med. 2026 Jan 1;394(1):13-26. doi: 10.1056/NEJMoa2512071. Epub 2025 Oct 19. PMID 41124220